CLINICAL TRIAL: NCT02232763
Title: A Prospective, Randomized, Cross-over Study Evaluating the Efficacy and Safety of Losartan in Pediatric Chronic Kidney Disease With Tubular Proteinuria
Brief Title: Efficacy and Safety of Losartan in Pediatric Chronic Kidney Disease With Tubular Proteinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Losartan_tubularPU_2014
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2017-07

CONDITIONS: Proteinuria
Keywords: Losartan; children; proteinuria
MeSH Terms: conditions — Proteinuria | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Losartan (Experimental): 12 weeks of losartan or placebo with crossover to the other
  Interventions: Drug: Losartan
- Placebo (Experimental): 12 weeks of losartan or placebo with crossover to the other
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — 12 weeks of losartan or placebo with crossover to the other
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — 12 weeks of losartan or placebo with crossover to the other
  Arms: Placebo

SUMMARY:
The investigators hypothesize that using Losartan would help decrease proteinuria in pediatric chronic kidney disease with tubular proteinuria.

DETAILED DESCRIPTION:
Children with tubular proteinuria (urine protein to creatinine ratio > 0.3 mg/mg) were randomly assigned in 1:1 ratio to losartan or placebo treatment for 12 weeks, then crossed over to the opposite intervention for another three months after a washout period of 2 weeks. The primary outcome is the change in urinary protein-creatinine ratio from baseline to the end of 12 weeks. Efficacy of losartan in children with CKD with tubular proteinuria was also investigated with additional retrospective review of medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2years or older and younger than 18 years
* estimated GFR ≥ 30mL/min/m^2
* Mean urinary protein-creatinine ratio > 0.3 g/g from three first-morning spot urine collections
* Renal hypoplasia/dysplasia, Reflux nephropathy, Polycystic kidney disease, Lowe syndrome, Dent disease, Tubulointerstitial nephritis, Nephronophthisis/Medullary cystic disease, Obstructive uropathy(including PUV, UPJ obstruction, UVJ obstruction)

Exclusion Criteria:

* hypertension
* under dialysis or organ transplanted
* bilateral renal artery stenosis or primary hyperaldosteronism
* pregnant or nursing

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
the change in urinary protein-creatinine ratio from baseline to the end of 12 weeks | 12 weeks
  Change in urinary protein excretion, determined as urinary Protein-creatinine ratio compared to baseline, after 12 weeks of treatment

SECONDARY OUTCOMES:
the change in urinary albumin-creatinine ratio from baseline to the end of study | 12 weeks
  Change in urinary albumin excretion, determined as urinary albumin-creatinine ratio compared to baseline, after 12 weeks of treatment
the proportion of patients wifh more than 50% decrease of urinary protein-creatinine ratio | 12 weeks
  number of patients with wifh more than 50% decrease of urinary protein-creatinine ratio compared to baseline, after 12 weeks of treatment
the change in urinary beta2-microglobulin-creatinine ratio from baseline to the end of study | 12 weeks
  Change in urinary beta2-microglobulin--creatinine ratio compared to baseline, after 12 weeks of treatment
the change in urinary NAG-creatinine ratio from baseline to the end of study | 12 weeks
  Change in urinary NAG-creatinine ratio compared to baseline, after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hee Gyung Kang, Ph.D, Study Chair — Seoul National University Children's Hospital Departments of Pediatrics
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea